CLINICAL TRIAL: NCT07282041
Title: Role of Glucagon-like Peptide 1 Receptor Agonist (GLP1 RA) Dulaglutide on Cerebral Hemodynamics In Patients With Severe and symptomAtic steNosis of inTracranial Internal Carotid Artery or Middle Cerebral Artery With Impaired Cerebral Vasodilatory Reserve- an Open-label Randomised Clinical Trial (RADIANT)
Brief Title: Role of GLP1 RA Dulaglutide on Severe Intracranial Atherosclerosis
Acronym: RADIANT
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National University of Singapore (Other)
Responsible Party: Principal Investigator, VIJAY KUMAR SHARMA, Associate Professor, National University of Singapore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RADIANT01
Record Dates: First submitted 2025-12-02; First posted 2025-12-15 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Intracranial Atherosclerosis; Stroke, Ischemic
MeSH Terms: conditions — Intracranial Arteriosclerosis; Ischemic Stroke | interventions — dulaglutide

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial
Who Masked: Outcomes Assessor
Masking Description: Study end-points would be assessed by independent investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dulaglutide (Experimental): Study participants would receive standard medical therapy plus Dulaglutide
  Interventions: Drug: Dulaglutide
- Standard medical therapy (No Intervention): Study participants would receive standard medical therapy

INTERVENTIONS:
Drug: Dulaglutide — Study participants would be randomised (1:1) to receive standard medical therapy or Dulaglutide plus standard medical therapy
  Arms: Dulaglutide

SUMMARY:
One important mechanism of action of GLP1 RA is the improvement in endothelial function, which may be evaluated by the assessment of cerebral vasodilatory reserve (CVR) in patients with severe ICAD. The investigators believe that GLP1 RA would be beneficial for patients with severe ICAD and lead to an improvement in cerebral vasodilatory reserve (CVR) in patients with severe and recently symptomatic stenosis of intracranial carotid artery (ICA) or middle cerebral artery (MCA).

In this open label randomised clinical trial, patients with recently symptomatic and severe stenosis of intracranial carotid artery (ICA) or middle cerebral artery (MCA) with impaired cerebral vasodilatory reserve (CVR) will be included. CVR will be measured with transcranial Doppler (TCD) breath holding index and acetazolamide-challenged single photon emission computed tomography (SPECT). Patients meeting the eligibility criteria would be randomised to receive best medical therapy (according to the international guidelines and institutional practices) or Dulaglutide subcutaneous injection (0.75mg and titrating to 1.5mg, if indicated) once a week, in addition to the best medical therapy. CVR will be measured again at the completion of 1 year. MRI of the brain will be repeated to evaluate any new ischaemic brain lesions. All patients would be followed up for two years for cerebral ischaemic events.

The investigators hypothesize that addition of GLP1 RA therapy would lead to a reduction of at least 4 units in CVR on SPECT as compared to best medical therapy.

DETAILED DESCRIPTION:
1. BACKGROUND AND RATIONALE Intracranial large artery atherosclerotic disease (ICAD) is widely prevalent among Asians. The risk of subsequent cerebral ischaemic episodes in ICAD ranges from 10-30% within 1-year despite current best medical treatment, being higher in patients with severe stenosis.

   1.1 General Introduction Recent glucose-lowering cardiovascular outcomes trials suggested that glucagon-like peptide 1 receptor agonist (GLP1 RA) reduced major adverse cardiovascular events (CVOTs), including non-fatal stroke. However, the mechanism(s) by which these agents reduce stroke remains unclear.

   1.2 Rationale and justification for the Study One important mechanism of action of GLP1 RA is the improvement in endothelial function, which may be evaluated by the assessment of cerebral vasodilatory reserve (CVR) in patients with severe ICAD. We believe that GLP1 RA would be beneficial for patients with severe ICAD and lead to an improvement in cerebral vasodilatory reserve (CVR) in patients with severe and recently symptomatic stenosis of intracranial carotid artery (ICA) or middle cerebral artery (MCA).

   In this open label randomised clinical trial, patients with recently symptomatic and severe stenosis of intracranial carotid artery (ICA) or middle cerebral artery (MCA) with impaired cerebral vasodilatory reserve (CVR) will be included. CVR will be measured with transcranial Doppler (TCD) breath holding index and acetazolamide-challenged single photon emission computed tomography (SPECT). Patients meeting the eligibility criteria would be randomised to receive best medical therapy (according to the international guidelines and institutional practices) or Dulaglutide subcutaneous injection (0.75mg and titrating to 1.5mg, if indicated) once a week, in addition to the best medical therapy. CVR will be measured again at the completion of 1 year. MRI of the brain will be repeated to evaluate any new ischaemic brain lesions. All patients would be followed up for two years for cerebral ischaemic events.

   The investigators hypothesize that addition of GLP1 RA therapy would lead to a reduction of at least 4 units in CVR on SPECT as compared to best medical therapy.
   1. Rationale for the Study Purpose GLP1 receptor agonists (GLP1 RA) beyond glucose lowering Glucagon-like peptide 1 (GLP1) was discovered in 1987. GLP1 enhances release of insulin in response to ingestion of glucose, known as incretin effect. In addition to the insulin release, GLP1 exerts other effects that improve glucose metabolism. Also, GLP1 delays gastric emptying and increase satiety, making it an ideal target for diabetes and obesity treatment. People with type 2 diabetes mellitus (T2DM) often have reduced incretin effect. The first GLP1 receptor agonist (GLP1 RA) exenatide, was approved in 2005 to treat T2DM. Since then, several GLP1 RAs have been developed. Most of the GLP1 RAs are given via subcutaneous injection-semaglutide, albiglutide, and dulaglutide administered via once-weekly injections, an attractive option for patients with T2DM, providing convenience and compliance.

      GLP1 RA were not primarily tested for their effect on reducing stroke risk! In 2008, FDA mandated that all trials related to the use of newer diabetes drugs report cardiovascular outcomes trials (CVOTs), after the experience from ACCORD (Action to Control Cardiovascular Risk in Diabetes) trial, which reported higher mortality due to cardiovascular causes with intensive glycaemic control.

      The mandated CVOTs for the new diabetes drugs are hailed as transformative as the CVOTs revealed cardioprotective effects of GLP1 RAs that shifted the treatment paradigm of T2DM.

      GLP1 RAs reduced MACE (major adverse cardiovascular events) which consists of cardiovascular death, non-fatal myocardial infarction, and non-fatal stroke. Interestingly, the reduction in the MACE was driven by the reduction in the non-fatal stroke, in particular for the once-weekly injection GLP1 RAs, Semaglutide and Dulaglutide. However, these trials reported stroke as a composite of all subtypes of strokes.

      There was no information about the presence of ICAD in GLP1 RA trials. While a better control of DM may lead to reduced cerebral ischaemia in patients with small vessel disease (lacunar strokes), whether patients with ICAD also derived similar benefit remains unknown. Since one of the important effects of GLP1 RA is through improvement of endothelial function, the investigators strongly believe that patients with severe ICAD (with impaired CVR-thus presumed endothelial dysfunction) may derive a preferential benefit in preventing cerebral ischaemic episodes.

      GLP1 RA and its potential in stroke prevention in ICAD Diabetic patients have a disproportionately higher risk of stroke and post-stroke mortality and morbidities (poor functional outcomes and high risk of recurrences). The findings of GLP1 RAs in reducing non-fatal stroke in several trials and meta-analyses provide the strong motivation to examine the hypothesis that GLP1 RA may reduce the risk of stroke among patients with ICAD. If proven, GLP1 RA treatment will bridge the clinical gap and change the treatment guidelines for managing high-risk patients.
   2. Rationale for Study Population Our target population is patients with recently symptomatic and severe stenosis of intracranial ICA or MCA, with impaired vasodilatory reserve on acetazolamide challenge SPECT. All patients will undergo similar evaluations at similar time-points.
   3. Rationale for Study Design One important mechanism of action of GLP1 RA is the improvement in endothelial function, which may be evaluated by the assessment of cerebral vasodilatory reserve (CVR) in patients with severe ICAD. The investigators believe that GLP1 RA would be beneficial for patients with severe ICAD and lead to an improvement in cerebral vasodilatory reserve (CVR) in patients with severe and recently symptomatic stenosis of intracranial carotid (ICA) or middle cerebral artery (MCA).

   In this open label randomised clinical trial, patients with recently symptomatic and severe stenosis of ICA or MCA with impaired CVR will be included. CVR will be measured with TCD breath holding index and acetazolamide-challenged SPECT. Patients meeting the eligibility criteria would be randomised to receive best medical therapy (according to the international guidelines and institutional practices) or Dulaglutide subcutaneous injection (0.75mg and titrating to 1.5mg) once a week, in addition to the best medical therapy. CVR will be measured again at the completion of 1 year. MRI of the brain will be repeated to evaluate any new ischaemic brain lesions. All patients would be followed up for two years for cerebral ischaemic events.

   The investigators hypothesize that addition of GLP1 RA therapy would lead to a reduction of at least 4 units in CVR on SPECT as compared to best medical therapy.
2. HYPOTHESIS AND OBJECTIVES

2.1 Primary Objectives- To evaluate whether GLP1 RA (Dulaglutide) therapy would lead to an improvement in cerebral vasodilatory reserve (CVR) by at least 4 points in patients with recently symptomatic and severe stenosis of ICA or MCA.

2.2 Secondary Objectives i) To evaluate the impact of GLP1 agonist (Dulaglutide) therapy on recurrence of cerebral ischaemic event in patients with recently symptomatic and severe stenosis of intracranial internal carotid artery (ICA) or middle cerebral artery (MCA) within 1 year (to evaluate treatment effect during therapy).

ii) To evaluate whether GLP1 agonist (Dulaglutide) therapy would reduce myocardial infarction (MI), all-cause mortality, and major adverse cardiovascular events (MACE, including cardiovascular death, nonfatal MI, and/or nonfatal ischaemic stroke) within 2 years (to evaluate sustained benefits).

2.4 Potential Risks and benefits:

1. End Points - Efficacy

   Primary endpoint:

   Change in CVR on acetazolamide SPECT at the end of the treatment from baseline.

   Secondary endpoints:

   A. Occurrence of TIA or stroke in the territory of the affected intracranial artery within 1-year of follow up.

   B. TIA or stroke or myocardial infarction (MI), all-cause mortality, and major adverse cardiovascular events (MACE, including cardiovascular death, nonfatal MI, and/or nonfatal ischaemic stroke) within 2-years follow up.
2. End Points - Safety For patients randomised to receive Dulaglutide, the investigators will record if any adverse reactions (pain at injection site, nausea, vomiting, stomach pain, indigestion, diarrhoea, loss of appetite, episodes of hypoglycemia or skin rashes etc).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 21 - 80 years old inclusive,
* Able to provide consent,
* Score 3 or less on the Modified Rankin Score (mRS),
* Patients with TIA or mild stroke with severe stenosis of intracranial ICA or MCA and impaired CVR within previous 3-months of acute stroke or TIA

Exclusion Criteria:

* Chronic kidney disease stage 5 (eGFR<15 mL/min) or on dialysis,
* Cancer diagnosed within past 3 years,
* Currently being planned for coronary or carotid artery revascularization,
* History of previous pancreatitis,
* History of medullary thyroid cancer,
* Atrial fibrillation,
* Any other condition likely to limit protocol compliance (judged by investigator).
* For diabetic patients, patients should not be on Sodium-glucose cotransporter 2 (SGLT2) inhibitor or pioglitazone during the duration of the study, unless these drugs can be stopped without affecting participants' medical condition. For those on Dipeptidyl peptidase-4 (DPP IV) inhibitor, this agent will be discontinued if the patient is randomised to the intervention group.
* Known allergies to Acetazolamide.
* Women who are pregnant or breastfeeding.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2025-12-17 (Actual); Primary Completion 2030-12-01 (Estimated); Study Completion 2030-12-01 (Estimated)

PRIMARY OUTCOMES:
To evaluate whether GLP1 RA (Dulaglutide) therapy would improveme cerebral vasodilatory reserve by at least 4 points in patients with severe stenosis of ICA or MCA | within 1 year
  To evaluate whether GLP1 RA (Dulaglutide) therapy would lead to an improvement in cerebral vasodilatory reserve (CVR) by at least 4 points in patients with recently symptomatic and severe stenosis of ICA or MCA.

SECONDARY OUTCOMES:
To evaluate the impact of Dulaglutide on recurrence of cerebral ischaemic event within 1 year. | within 1year
  To evaluate the impact of GLP1 agonist (Dulaglutide) therapy on recurrence of cerebral ischaemic event in patients with recently symptomatic and severe stenosis of intracranial internal carotid artery (ICA) or middle cerebral artery (MCA) within 1 year (to evaluate treatment effect during therapy).
To evaluate whether Dulaglutide would reduce MACE within 2 years | within 2 years
  To evaluate whether GLP1 agonist (Dulaglutide) therapy would reduce myocardial infarction (MI), all-cause mortality, and major adverse cardiovascular events (MACE, including cardiovascular death, nonfatal MI, and/or nonfatal ischaemic stroke) within 2 years (to evaluate sustained benefits).

CONTACTS AND LOCATIONS:
Overall Officials: vijay K sharma, MD, Principal Investigator — National University of Singapore
Locations (1):
- National University Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
Upon completion of the study, the team would decide about sharing anonymised patient data with other researchers